CLINICAL TRIAL: NCT05769491
Title: Investigation of Patterns in Clinical Trial Experiences by Patients Participating in Triple Negative Breast Cancer Clinical Trials
Brief Title: Looking At Triple Negative Breast Cancer Patient Experience Patterns in Medical Trials
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 84434789
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Triple Negative Breast Cancer; Breast Cancer
Keywords: triple negative breast cancer; breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical trials can sometimes favor certain demographic groups. Additionally, there is limited research that delves into the factors that influence participation in clinical trials, both positive and negative.

The goal is to identify the obstacles and challenges that prevent participation in Triple Negative Breast Cancer clinical trials, as well as the reasons for withdrawal or discontinuation.

The insights gained from this study will ultimately benefit those with Triple Negative Breast Cancer who may be invited to participate in clinical research in the years to come.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Willing and able to comply with scheduled visits, treatment schedule, laboratory tests and other requirements of the study.
* Capable of giving signed informed consent, which includes compliance with requirements and restrictions listed in the informed consent form (ICF) and in the protocol

Exclusion Criteria:

* Pregnant or lactating woman
* Any mental or medical condition that prevents the patient from giving informed consent or participating in the trial
* Inability to perform regular electronic reporting

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Triple negative breast cancer patients who are actively considering participating in an observational medical study, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Number of triple negative breast cancer patients who decide to enroll in a clinical study | 3 months
Rate of triple negative breast cancer patients who remain in a clinical study to completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shao Z, Chaudhri S, Guo M, Zhang L, Rea D. Neoadjuvant Chemotherapy in Triple Negative Breast Cancer: An Observational Study. Oncol Res. 2016;23(6):291-302. doi: 10.3727/096504016X14562725373879. PMID 27131315
- [Background] Wu B, Sun C, Sun X, Li X. The effect of chemotherapy on survival in oldest old patients with nonmetastatic triple negative breast cancer: A populationbased observational study. J Clin Pharm Ther. 2022 Nov;47(11):1826-1836. doi: 10.1111/jcpt.13776. Epub 2022 Sep 29. PMID 36175133
- [Background] Costa REARD, Oliveira FTR, Araujo ALN, Vieira SC. Prognostic factors in triple-negative breast cancer: a retrospective cohort. Rev Assoc Med Bras (1992). 2021 Jul;67(7):950-957. doi: 10.1590/1806-9282.20210249. PMID 34817505

DOCUMENTS (1):
  • Informed Consent Form (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/91/NCT05769491/ICF_000.pdf